CLINICAL TRIAL: NCT03853395
Title: BIOmarker-guided Treatment Decisions in Psoriatic and Rheumatoid Arthritis: a Feasibility Study
Brief Title: BIOTIPRA: BIOmarker-guided Treatment Decisions in Psoriatic and Rheumatoid Arthritis
Acronym: BIOTIPRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr. James Bluett, Chief Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHS001481
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator): Participants on this arm of the study will provide trough blood samples and complete participant questionnaires. Their research teams will return clinical information about them to the University of Manchester. Clinicians for this group of participants will not receive blood results (about drug levels or anti-drug antibodies) or treatment advice from the University of Manchester about their participant.
  Interventions: Diagnostic Test: Tests for drug levels and anti-drug antibodies
- Experimental Arm (Experimental): Participants on this arm of the study will provide trough blood samples and complete participant questionnaires. Their research teams will return clinical information about them to the University of Manchester. Clinicians for this group of participants will receive blood results (about drug levels or anti-drug antibodies) or treatment advice from the University of Manchester about their participant. They will be able to act accordingly.
  Interventions: Diagnostic Test: Tests for drug levels and anti-drug antibodies

INTERVENTIONS:
Diagnostic Test: Tests for drug levels and anti-drug antibodies — Measurement of drug levels and anti-drug antibodies will be undertaken using commercially available enzyme-linked immunosorbent assays (ELISAs) and/or radioimmunoassays

SUMMARY:
TNFi drugs remain the most prescribed first-line biologics for patients with rheumatoid arthritis (RA). However, up to 40% of RA patients fail to respond to TNFi treatment. One explanation of non-response is the development of anti-drug antibodies and low drug levels.

Studies have consistently shown that:

1. Serum drug levels of monoclonal antibodies (such as adalimumab, certolizumab, infliximab) and the presence of anti-drug antibodies in samples taken at 3 and 6 months correlate with subsequent response at 12 months.
2. Non-responders and those who develop anti-drug antibodies are less likely to receive concomitant methotrexate or, if they do receive it, are on lower doses than responder groups.

However, it has not been proven that knowing that a patient had low drug levels or anti-drug antibodies would have improved the outcome; neither has it been shown that introducing or increasing the dose of methotrexate would reduce the formation of anti-drug antibodies, thereby improving outcome.

Observational data has revealed that RA non-responders, who exhibit adequate serum drug levels and no detectable anti-drug antibodies, have lower probability of response to another agent with the same mechanism of action (MOA), and may benefit in switching to a drug with a different MOA (12). RA non-responders, who have low detectable serum trough levels and detectable anti-drug antibodies, may benefit in switching to a less immunogenic drug (13, 14). These patients may have a predisposition of developing immunogenicity against the introduced foreign protein (12). Neutralising anti-drug antibodies against the TNFi etanercept or the T-cell co-stimulation inhibitor abatacept have not been detected (10, 12, 15). Furthermore whilst the use and dose of methotrexate at initiation of TNFi, has been associated with lower levels of anti-drug antibodies in our work and others (10, 16), it is not known if increasing the MTX dose once immunogenicity has developed reduces anti-drug antibodies and leads to improved treatment response.

Whilst algorithms have been proposed based on these tests (4, 17, 18), they have not been confirmed in a randomised controlled trial setting to show that the intervention (testing) is effective. Based on our preliminary work in an observational dataset, this feasibility study will allow us to design a definitive study to answer the important issue of whether pharmacological testing can be utilised as robust biomarkers to optimise future patient outcomes.

The next essential step, therefore, is to prove that introducing these tests improves clinical outcome. It is very important to do so because some clinicians are already requesting that their immunology laboratories introduce such tests; yet the tests themselves are expensive and have not yet shown efficacy (19). Conducting a clinical feasibility trial is one of the essential first steps in development of a full clinical trial to undertake process evaluation and assess the proposed study design, required number of participants and ensure optimum project completion.

The proposed trial is a clinical feasibility trial with the aim to ensure a realistic assessment and capability to conduct the full clinical trial. Participants with RA, commencing adalimumab or certolizumab will be randomised to determine whether providing test results on adalimumab/certolizumab drug levels and anti-drug antibodies at 4 weeks, 3 and 6 months to clinicians caring for patients with RA (n=15 patients) starting on treatment with adalimumab/certolizumab, improves the course of disease activity, compared to standard care (n=15 patients). Clinicians will be provided with feedback and a treatment algorithm. The feasibility of the study will be assessed by a number of factors including evaluation of recruitment, attrition, data completeness and process evaluation. The results will be used to inform the number of participants required to fully evaluate the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RA about to start therapy with adalimumab or certolizumab
2. Age 18 and over, male or female
3. Willing to take part in the study
4. Patients who consent to take part in the BRAGGSS study

Exclusion Criteria:

1. Patients unwilling or unable to take part in the study
2. Pregnant women or nursing (breast feeding) mothers.
3. Planned pregnancy within next 12 months.
4. Scheduled surgery in the next 12 months or other pre-planned reasons for treatment discontinuation in the next 12 months.
5. Contraindication to adalimumab or certolizumab according to the summary of product characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
1. Power for full randomised controlled trial: Change in Disease Activity Score (DAS)-28 over 12 months | through study completion, an average of 1 year
2. Process evaluation: Patient/care-giver opinion of measuring adalimumab/certolizumab drug levels and anti-drug antibodies with feedback using a specially adapted questionnaire | through study completion, an average of 1 year
3. Process evaluation: Patient and care-giver opinion of process of research, including outcome measures measured by a specially adapted questionnaire | through study completion, an average of 1 year
4. Process evaluation: fidelity and quality of trial implementation and success of recruitment strategy | through study completion, an average of 1 year
  A mixed-methods process evaluation will explore the fidelity and quality of implementation through evaluation of missing and non-missing responses. To inform the decision to proceed to a full clinical trial evaluation will take place measuring intervention fidelity; recruitment time; uptake; patient acceptability; withdrawal rate; effect size; affordability; study period required; time required for drug measurement and patient perspectives.

SECONDARY OUTCOMES:
1. Change in Health Assessment Questionnaire (HAQ) measurement | through study completion, an average of 1 year
2. Change in Short Form 36 (SF-36) | through study completion, an average of 1 year
3. Change in SF-36 vitality subscale | through study completion, an average of 1 year
4. Health Assessment Questionnaire Disability Index at 12 months | through study completion, an average of 1 year
5. Change in pain Visual Analog Scale (VAS) | through study completion, an average of 1 year
6. Percentage of patients with increase in MTX dose | through study completion, an average of 1 year
7. Percentage of patients with reduction of anti-drug antibody formation | through study completion, an average of 1 year
8. Percentage of patients who stop TNFi and experience disease flare within 12 months of recruitment | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Centre for Musculoskeletal Research, Manchester, England
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Midlands Partnership NHS Foundation Trust, Stafford, Staffordshire
  - Leicester Royal Infirmary, Leicester
  - Homerton University Hospital NHS Foundation Trust, London
  - Manchester University Hospitals NHS Foundation Trust, Manchester
  - Northern Care Alliance NHS Group, Manchester
  - Torbay and South Devon NHS Foundation Trust, Torquay
  - Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
No person identifiable information (PII, as defined by the GDPR) will be made available to other researchers. Other bone fide may access other information upon request to Dr. James Bluett.